CLINICAL TRIAL: NCT07253727
Title: The LUCENT Study - LUng Lesion Assessment Via BF-UCP190F for Central and Extended Nodal Targeting
Acronym: LUCENT
Status: Not yet recruiting | Type: Observational
Sponsor: Olympus Europe SE & Co. KG (Industry)
Collaborators: Heidelberg University (Other); Lung Clinic Hemer (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-02
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Bronchoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indicated for bronchoscopy
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — no intervention, only observational

SUMMARY:
The Olympus BF-UCP190F bronchoscope combines the reach of a thinner bronchoscope with the benefit of real-time ultrasound, enabling direct lesion visualization and sampling deeper into the lung. Following promising first-in-human data, the LUCENT study aims to evaluate the utility feasibility, effectiveness and safety of this device in a multicenter setting, generating real-world evidence to inform broader adoption in global markets.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. ≥18 years of age.
3. The target lesion(s) must be located within the inner and middle two-thirds of the lung, as determined prospectively using the Software-Assisted Method (SAM). To ensure accurate localization, SAM applies anatomical measurements to classify lesions as inner, middle, or outer third of the lung. The lesion must contact the border of the inner two-thirds region; lesions fully outside this region will be excluded from the study cohort. In addition, the lesion must be located at least two airway generations distal to the main carina, as confirmed radiographically by the bronchoscopist
4. Target lesion: nodule ≥ 10mm or lymph node ≥ 5mm.
5. Target lesion location documented on CT or PET report.
6. Indicated for bronchoscopy.
7. Bronchoscopic procedure scheduled within 30 days of the CT or PET report.
8. Patient qualifies for a procedure using the BF-UCP190F bronchoscope and the ViziShot 2 25 needle based upon the approved indications for use for those devices.

Exclusion Criteria:

1. Concurrently participating in another competing clinical study.
2. Unwilling or unable to return for follow-up, e.g., plans for relocation, unsuitable transportation.
3. Patient not suitable for flexible bronchoscopy as determined by the treating physician prior to the procedure.
4. Currently on anticoagulation that cannot be paused, or a coagulation disorder that, in the opinion of the investigator, would pose an increased risk of bleeding.
5. Intraprocedural identification of intrinsic and endoscopically visualized endobronchial lesion for which adequate biopsy can be obtained via endobronchial biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indicated for bronchoscopy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Ability to visualize and sample a priori defined lesion in the inner or middle third of the lung with BF-UCP190F. | Index Procedure
  The primary endpoint-the proportion of a priori defined inner/middle-third lesions visualized and sampled using the BF-UCP190F-will be summarized using descriptive statistics, including frequency and percentage with 95% confidence intervals.

IPD SHARING:
Plan to Share IPD: No